CLINICAL TRIAL: NCT02330510
Title: Amyloid and Glucose PET Imaging in Alzheimer and Vascular Cognitive Impairment Patients With Significant White Matter Disease
Acronym: MITNEC C6
Status: Completed | Type: Observational
Sponsor: Dr. Sandra E Black (Other)
Responsible Party: Sponsor-Investigator, Dr. Sandra E Black, Principal Investigator, Sunnybrook Health Sciences Centre
Organization: Sunnybrook Health Sciences Centre (Other)
Other Study IDs: Ml1-112246
Record Dates: First submitted 2014-06-27; First posted 2015-01-05 (Estimated); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Alzheimer's Disease; Small Vessel Disease White Matter Hyperintensities Subtype; Vascular Cognitive Impairment
Keywords: Alzheimer's Disease; White Matter Hyperintensities; Vascular Cognitive Impairment; Amyloid Imaging; Transient Ischemic Attack
MeSH Terms: conditions — Alzheimer Disease; Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood will be collected to better understand the possible contribution of genetics to white matter disease. DNA will be extracted from blood samples to assess the Apolipoprotein (ApoE) gene type, as ApoE e4 genotype may influence the rate of disease progression.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Alzheimer's Disease: Individuals with early Alzheimer's Disease (AD) or amnestic or multi-domain Mild Cognitive Impairment who have extensive Periventricular White Matter Hyperintensities
- Transient Ischemic Attack/Mild Subcortical Stroke: Individuals who have had a mild subcortical stroke or a Transient Ischemic Attack (TIA) with extensive Periventricular White Matter Hyperintensities in the absence of cortical infarcts

SUMMARY:
The prevalence of both Alzheimer's Disease (AD) and stroke doubles each decade over 65 years old. Both are major causes of dementia, currently estimated to affect 46 million people worldwide. The current costs globally are $818 billion. Additionally, in population studies elders over 65 years, "covert" cerebral small vessel disease appears on MRI scans as silent lacunar infarcts in 25% as Microbleeds in 10%, and as focal or diffuse 'incidental' white matter disease (WMD) in 95%. WMD is extensive in 20%, with a clinical threshold effect around 10cc2. Small vessel disease is even more common in dementia, often coexisting with AD and independently contributing to cognitive decline and progression to dementia. Longitudinal imaging using cerebral amyloid labeling opens a new opportunity to understand the additive/interactive effects of small vessel disease and AD.

The design of this study includes recruitment of two cohorts, including Mild Cognitive Impairment (MCI) and/or early Alzheimer Disease subjects from memory clinics and subjects with strokes/TIA from stroke prevention clinics. Inclusion criteria include the presence of moderate/extensive white matter disease, eg. Fazekas score of 2 (with confluent peri-ventricular hyperintensities) or Fazekas score of 3, as determined by previous MR or CT, > 60 years of age, Mini-Mental Status Exam (MMSE) scores ≥ 20. Subjects will undergo 3T structural MRI (including T1, PD/T2, FLAIR, GRE, DTI, ASL, and resting state fMRI), glucose PET, amyloid PET (using AV-45 florbetapir) and neuropsychological testing, as well as blood sampling. Repeat MR and PET/CT imaging and neuropsychological testing will be conducted at 24 months. The follow up assessments can also be completed at either year 1 or year 3 or Year 4 depending on the availability of study participants. The imaging portion is designed to closely parallel the Alzheimer's Disease Neuroimaging Initiative (ADNI) in order to benefit from the availability of both cognitively normal controls (NC), MCI and Alzheimer's disease subjects with minimal WMD.

DETAILED DESCRIPTION:
This study will be a multi-center trial to be conducted in centers across Canada and approximately 80 patients will be enrolled. Participants will be recruited from both stroke prevention (N=40) and memory clinics (N=40). For comparison, we will access the publically-available data using a very similar protocol being collected from normal controls (N=250), MCI (N=250 early MCI, N=150 late MCI) and AD patients (N=150) without significant white matter disease, who are participating in the Alzheimer's Disease Neuroimaging Initiative (ADNI-GO and ADNI 2, N=800), to choose representative samples for comparison to those with scores ≤ 1 who represent the non-white matter disease group.

Three imaging modalities will be used with each participant. 3 Telsa MRI scans will be acquired, using an ADNI based protocol, except for the addition of a PD/T2 interleved sequence. Participants will also undergo 18-fluoro PET with the AVID-45 ligand and 18-fluorodeoxyglucose PET using the ADNI protocols.

The primary objectives are to characterize at baseline and 2-year follow-up in patients with significant Periventricular White Matter Hyperintensities (pvWMH), presenting as transient cerebrovascular events or memory problems, patterns of: 1. Uptake of amyloid on Florbetapir F-18 PET/CT 2. Glucose uptake on 18F-FDG PET/CT 3. Volumetric measures of brain structure on MRI imaging 4. Performance on standard neuropsychological assessments, activities of daily living and gait speed.

Secondary objectives are to: 1. Compare the relationship between amyloid brain uptake, pvWMH volumes, and cognitive scores in patients with significant pvWMH and a control group of individuals that are cognitively normal, MCI or AD, with mild pvWMH, identified from the ADNI database. 2. Examine the relationship between amyloid uptake, ApoE e4 genotype, and structural MRI volumes in patients with a high burden of pvWMH. 3. Evaluate the utility of baseline brain amyloid to predict cognitive decline and increases in pvWMH volume at 2 years follow up. 4. Evaluate the safety of a single intravenous dose of Florbetapir F 18 Injection (370 MBq +/- 10%) in subjects with significant pvWMH.

ELIGIBILITY:
Eligible subjects must meet the following criteria before they are enrolled into the study:

1. Patients with early AD or amnestic, non-amnestic single or multi-domain MCI who have confluent pvWMH; recruited from memory clinics. Or Patients who have had a minor stroke (e.g. subcortical lacunar infarct ≤1.5cm) or a TIA with confluent pvWMH; recruited from stroke prevention clinics.
2. Age ≥ 60
3. Patients who have provided written informed consent
4. Patients with greater than 8 years of education
5. Patients with an expected survival of greater than 2 years
6. Patients that are sufficient fluency in French or English for cognitive testing
7. Patients with a Mini-Mental State Exam score of (MMSE) ≥ 20
8. Patients with pvWMH score on CT or MRI of ≥2 on the periventricular Fazekas scale 31 NOTE: Fazekas 2 patients can be included if they have bilateral posterior or anterior periventricular caps extending only 10mm from the ventricle (i.e. halfway into the surrounding white matter vs extending out to most of the surrounding white matter required for Fazekas 3)

Exclusion Criteria:

1. Subject meeting any one of the following criteria are not eligible for the the study:
2. Patients with cortical or non-lacunar infarct on imaging
3. Patients with persisting hemiparesis after a motor stroke, leg strength <4/5 on the Medical Research Council (MRC) scale; significant cerebellar ataxia
4. Patients with contraindications to 3T MRI
5. Patients with major psychiatric disorder during the preceding 5 years
6. History of substance abuse within the past 2 years
7. Serious/chronic systemic or neurological illness (other than AD) such as Parkinson's disease, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma followed by persistent neurologic deficits or known structural brain abnormalities
8. Pain or sleep disorder that could interfere with testing
9. Claustrophobia
10. Patients that have received radiation therapy to the head or neck or have been in another research study involving radiation
11. Patients who are unable or unwilling to comply with protocol requirements or deemed by the investigator to be unfit for the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two groups of patients will participate in this study:
  1. Patients with early Alzheimer's Disease (AD) or amnestic or multi-domain Mild Cognitive Impairment who have extensive pvWMH; recruited from memory clinics (n= 40)
  2. Patients who have had a stroke or a Transient Ischemic Attack (TIA) with extensive pvWMH; recruited from stroke prevention clinics (n= 40)
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Change in F18 florbetapir SUVR over 2 years in patients with moderate-severe White Matter Hyperintensities, at baseline and 1 year follow-up brain uptake of Florbetapir F 18 | 24 months
  Standardized measures of F18 florbetapir brain uptake will be compared to baseline uptake patterns and prevalence of signal uptake in various areas

SECONDARY OUTCOMES:
Florbetapir F18 SUVR brain uptake, regional FDG metabolic measures and regional volutmetrics on MRI based volume including grey and white matter, small vessel disease, as well as regional cortical thickness measures. | 24 months
  Standardized measures of F18 florbetapir brain uptake will be correlated with posterior-cingulate and parietal-temporal metabolism. We will also correlate with hippocampal, ventricular and regional volumes and with cortical thickness, derived with Lesion Explorer enhancement
F18 florbetapir SUVR brain uptake, with Periventricular White Matter Hyperintensity volumes and cognitive scores. | 24 months
  The relationship between F18 florbetapir brain uptake, Periventricular White Matter Hyperintensity volumes, executive function and memory scores, in patients with significant pvWMH, accounting for relevant co-variates (age, education), using multivariate analysis including Partial Least Squares (PLS).
F18 florbetapir brain SUVR uptake, Periventricular White Matter Hyperintensity volumes and cognitive scores in an age-matched group of normal controls, MCI and AD subjects with minimal or mild degrees of pvWMH. | 24 months
  Mutlivariate analysis will be used to carry out this analysis, including PLS
F18 florbetapir SUVR brain uptake, ApoE e4 genotype status, and White Matter Hyperintensity volumes in patients with a high burden of pvWMH. | 24 months
Baseline F18 florbetapir SUVR brain uptake, cognitive score decline and increase in White Matter Hyperintensity volume at 2 year follow up. | 24 months
Assess any adverse events or serious adverse events occurring with a a single intravenous dose of F18 florbetapir Injection (370 MBq +/- 10%) in subjects with significant pvWM | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Sandra E. Black, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (8):
- Canada (8):
  - University of Alberta Health Services, Calgary, Alberta
  - University of British Columbia Hospital, Vancouver, British Columbia
  - Hamilton General Hospital, Hamilton, Ontario
  - Parkwood Hospital St. Joseph's Health Care, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - CHU de Sherbrooke, Québec, Quebec
  - CHU de Quebec, Québec, Quebec

REFERENCES:
- [Derived] Xhima K, Ottoy J, Gibson E, Zukotynski K, Scott C, Feliciano GJ, Adamo S, Kuo PH, Borrie MJ, Chertkow H, Frayne R, Laforce R Jr, Noseworthy MD, Prato FS, Sahlas DJ, Smith EE, Sossi V, Thiel A, Soucy JP, Tardif JC, Goubran M, Black SE, Ramirez J; Medical Imaging Trials Network of Canada (MITNEC). Distinct spatial contributions of amyloid pathology and cerebral small vessel disease to hippocampal morphology. Alzheimers Dement. 2024 May;20(5):3687-3695. doi: 10.1002/alz.13791. Epub 2024 Apr 4. PMID 38574400
- [Derived] Boone L, Biparva M, Mojiri Forooshani P, Ramirez J, Masellis M, Bartha R, Symons S, Strother S, Black SE, Heyn C, Martel AL, Swartz RH, Goubran M. ROOD-MRI: Benchmarking the robustness of deep learning segmentation models to out-of-distribution and corrupted data in MRI. Neuroimage. 2023 Sep;278:120289. doi: 10.1016/j.neuroimage.2023.120289. Epub 2023 Jul 24. PMID 37495197
- [Derived] Ottoy J, Ozzoude M, Zukotynski K, Kang MS, Adamo S, Scott C, Ramirez J, Swardfager W, Lam B, Bhan A, Mojiri P, Kiss A, Strother S, Bocti C, Borrie M, Chertkow H, Frayne R, Hsiung R, Laforce RJ, Noseworthy MD, Prato FS, Sahlas DJ, Smith EE, Kuo PH, Chad JA, Pasternak O, Sossi V, Thiel A, Soucy JP, Tardif JC, Black SE, Goubran M; Medical Imaging Trials Network of Canada (MITNEC) and Alzheimer's Disease Neuroimaging Initiative (ADNI). Amyloid-PET of the white matter: Relationship to free water, fiber integrity, and cognition in patients with dementia and small vessel disease. J Cereb Blood Flow Metab. 2023 Jun;43(6):921-936. doi: 10.1177/0271678X231152001. Epub 2023 Jan 25. PMID 36695071
- [Derived] Ottoy J, Ozzoude M, Zukotynski K, Adamo S, Scott C, Gaudet V, Ramirez J, Swardfager W, Cogo-Moreira H, Lam B, Bhan A, Mojiri P, Kang MS, Rabin JS, Kiss A, Strother S, Bocti C, Borrie M, Chertkow H, Frayne R, Hsiung R, Laforce RJ, Noseworthy MD, Prato FS, Sahlas DJ, Smith EE, Kuo PH, Sossi V, Thiel A, Soucy JP, Tardif JC, Black SE, Goubran M; Medical Imaging Trial Network of Canada (MITNEC) and Alzheimer's Disease Neuroimaging Initiative (ADNI). Vascular burden and cognition: Mediating roles of neurodegeneration and amyloid PET. Alzheimers Dement. 2023 Apr;19(4):1503-1517. doi: 10.1002/alz.12750. Epub 2022 Sep 1. PMID 36047604
- [Derived] Mojiri Forooshani P, Biparva M, Ntiri EE, Ramirez J, Boone L, Holmes MF, Adamo S, Gao F, Ozzoude M, Scott CJM, Dowlatshahi D, Lawrence-Dewar JM, Kwan D, Lang AE, Marcotte K, Leonard C, Rochon E, Heyn C, Bartha R, Strother S, Tardif JC, Symons S, Masellis M, Swartz RH, Moody A, Black SE, Goubran M. Deep Bayesian networks for uncertainty estimation and adversarial resistance of white matter hyperintensity segmentation. Hum Brain Mapp. 2022 May;43(7):2089-2108. doi: 10.1002/hbm.25784. Epub 2022 Jan 28. PMID 35088930
- [Derived] Ntiri EE, Holmes MF, Forooshani PM, Ramirez J, Gao F, Ozzoude M, Adamo S, Scott CJM, Dowlatshahi D, Lawrence-Dewar JM, Kwan D, Lang AE, Symons S, Bartha R, Strother S, Tardif JC, Masellis M, Swartz RH, Moody A, Black SE, Goubran M. Improved Segmentation of the Intracranial and Ventricular Volumes in Populations with Cerebrovascular Lesions and Atrophy Using 3D CNNs. Neuroinformatics. 2021 Oct;19(4):597-618. doi: 10.1007/s12021-021-09510-1. Epub 2021 Feb 1. PMID 33527307